CLINICAL TRIAL: NCT06081049
Title: The COLchicine HEART Failure PRESERVED Trial (COLHEART-PRESERVED)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tor Biering-Sørensen (Other)
Responsible Party: Sponsor-Investigator, Tor Biering-Sørensen, Professor, Head of Center for Translational Cardiology and Pragmatic Randomized Trials, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COLHEART-PRESERVED
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Randomized Controlled Trial; Cardiovascular Diseases; Heart Diseases; Colchicine; Inflammation; Echocardiography; Hypertrophy, Left Ventricular; Ventricular Function, Left; Diastolic Dysfunction, Left Ventricular; Atrial Enlargement, Left; Quality of Life; Kansas City Cardiomyopathy Questionnaire
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Inflammation; Hypertrophy, Left Ventricular; Ventricular Dysfunction, Left | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Colchicine 0.5 mg once daily
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — 0.5 mg once daily
  Arms: Colchicine
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of colchicine on heart failure related health status, quality of life, and vascular and cardiac function in patients with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
The study is an investigator-initiated, prospective, randomized, double-blind, placebo-controlled study of the effects of colchicine in patients with HFpEF. The study population will consist of approx. 152 patients aged 40 years and above, who meet the criteria of HFpEF. Patients will be randomized to either low-dose colchicine treatment (0.5 mg once daily) or placebo and treatment will continue for 6 months. Patients will be assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ) and have echocardiography performed at baseline and after 6 months. Furthermore, the investigators will obtain office blood pressure, ECG, Myovista ECG, 6-minute walk test, pulse wave velocity (PWV), and blood samples at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≥ 45% judged by echocardiography during the screening epoch or within 6 months prior to screening visit
* Symptom(s) of heart failure for at least 30 days prior to screening visit and current symptoms of heart failure (NYHA functional class II-IV) at screening visit
* Objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of LV diastolic dysfunction/raised LV filling pressures (left atrial enlargement and/or left ventricular hypertrophy) judged by echocardiography at screening epoch or within 12 months prior to screening visit
* Raised pro-BNP ≥ 125 pg/ml (sinus rhythm) or ≥ 300 pg/ml (atrial fibrillation (AF)).
* Body Mass Index (BMI) < 40 kg/m2 at screening visit
* Female patients should either not be of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or of childbearing potential and practicing one of the following methods of contraception throughout the study and for 30 days after study completion: Hormonal contraception (oral contraceptives, contraceptive implant, injectable birth control, contraceptive patch, or vaginal ring) or intrauterine device
* Patients will have given written, informed consent and are able and willing to comply with the requirements of the study protocol

Exclusion Criteria:

* Colchicine treatment for another cause, e.g., gout
* Allergy/hypersensitivity to colchicine
* Uncontrolled hypertension (systolic BP >180 mmHg or diastolic BP >110 mmHg)
* History of malignancy of any organ system excluding a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma, localized prostate cancer and/or localized carcinoma in situ of the cervix
* Cirrhosis, chronic active hepatitis, or other severe hepatic disease
* Hemodialysis
* Estimated glomerular filtration rate (eGFR) < 35 mL/min/1.73 m2
* Systemic treatment with moderate or strong cytochrome P450 3A4 (CYP3A4) inhibitors or P-glycoprotein inhibitors
* Anemia, thrombocytopenia, or leucopenia defined as any of the following measurements within the last 3 months:

  * Hemoglobin < 7 mmol/L
  * Platelet count < 110 x 109/L
  * White blood cell count < 3.0 x 109/L
* Acute decompensated heart failure (hospitalization for heart failure within 7 days prior to screening visit)
* Acute coronary syndrome (including MI), cardiac surgery, other major cardiovascular surgery, ablation of atrial flutter/fibrillation, valve repair/replacement, implanted cardioverter defibrillator or urgent PCI within 3 months prior to screening visit or an elective PCI within 30 days prior to screening visit
* Planned coronary revascularization (percutaneous intervention or surgical), major cardiac surgery (coronary artery bypass grafting, valve repair/replacement, ventricular assist device, cardiac transplantation, or any other surgery requiring thoracotomy), CRT or ablation of atrial flutter/fibrillation during the trial
* Any clinical event within 6 months prior to screening visit that could have reduced LVEF (e.g., MI, CABG), unless echocardiographic measurement was performed after the event confirming LVEF ≥ 45%
* Stroke, transient ischemic attack, carotid surgery, or carotid angioplasty within 3 months prior to screening visit
* Previous cardiac transplantation, complex congenital heart disease or cardiac resynchronization therapy
* Heart failure due to any of the following: known infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac tamponade, known genetic hypertrophic cardiomyopathy, obstructive cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy or uncorrected severe/hemodynamically significant valvular heart disease
* Life threatening or uncontrolled dysrhythmia, including symptomatic or sustained ventricular tachycardia and AF or atrial flutter with a resting ventricular rate > 110 beats per minute
* Evidence of right-sided HF in the absence of left sided structural heart disease
* Probable alternative diagnosis that in the opinion of the investigator could account for the patient's HF symptoms (i.e., anemia, hypothyroidism, severe obesity)
* World Health Organization Group 1 pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease, including COPD (i.e., requiring home oxygen, chronic nebulizer therapy or chronic oral steroid therapy, or hospitalization for exacerbation of COPD requiring ventilatory assist within 12 months prior to enrollment)
* Female patients who are pregnant, lactating, or considering becoming pregnant during the study or for 6 months after study completion
* Significant drug or alcohol abuse during the last year
* Current use of or plans to initiate chronic systemic steroid therapy during the study (topical or inhaled steroids are allowed)
* Chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis) or chronic diarrhea
* Use of other investigational drugs within 30 days of the time of enrollment
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
* Life expectancy < 2 years at the screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in change in Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) at 6 months | 6 months
  The Kansas City Cardiomyopathy Questionnaire scores are scaled from 0-100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; 75 to 100; good to excellent.

SECONDARY OUTCOMES:
Between-group difference in change in Kansas City Cardiomyopathy Questionnaire Overall Summary Score (KCCQ-OS) at 6 months | 6 months
  The Kansas City Cardiomyopathy Questionnaire scores are scaled from 0-100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; 75 to 100; good to excellent.
Between-group difference in the proportion of patients with a ≥ 5-point increase in KCCQ-CS and KCCQ-OS at 6 months | 6 months
  The Kansas City Cardiomyopathy Questionnaire scores are scaled from 0-100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; 75 to 100; good to excellent.

OTHER OUTCOMES:
Between-group difference in change in office-measured systolic blood pressure at 6 months | 6 months
Between-group difference in change in office-measured diastolic blood pressure at 6 months | 6 months
Between-group difference in change in exercise capacity assessed by 6-minute walk test at 6 months | 6 months
Between-group difference in change in LV mass index assessed by echocardiography at 6 months | 6 months
Between-group difference in change in hs-CRP at 6 months | 6 months
Between-group difference in change in hs-TnI at 6 months | 6 months
Between-group difference in change in carotid-femoral pulse wave velocity at 6 months | 6 months
Between-group difference in change in office-measured pulse pressure at 6 months | 6 months
Between-group difference in change in central blood pressure at 6 months | 6 months
Between-group difference in change in augmentation index at 6 months | 6 months
Between-group difference in change in LV septal wall thickness assessed by echocardiography at 6 months | 6 months
Between-group difference in change in LV posterior wall thickness assessed by echocardiography at 6 months | 6 months
Between-group difference in change in LVEF assessed by echocardiography at 6 months | 6 months
Between-group difference in change in E/A ratio assessed by echocardiography at 6 months | 6 months
Between-group difference in change in e' assessed by tissue Doppler echocardiography at 6 months | 6 months
Between-group difference in change in early mitral inflow velocity to early diastolic mitral annular velocity (E/e' ratio) assessed by echocardiography at 6 months | 6 months
Between-group difference in change in early mitral inflow velocity to global diastolic strain rate (E/e'sr ratio) assessed by echocardiography at 6 months | 6 months
Between-group difference in change in left atrial volume (LAV) assessed by echocardiography at 6 months | 6 months
Between-group difference in change in global longitudinal strain (GLS) assessed by echocardiography at 6 months | 6 months
Between-group difference in change in TNF-α at 6 months | 6 months
Between-group difference in change in pro-BNP at 6 months | 6 months
Between-group difference in change in interleukin-1 beta at 6 months | 6 months
Between-group difference in change in interleukin-6 at 6 months | 6 months
Between-group difference in change in interleukin-10 at 6 months | 6 months
Between-group difference in change in interleukin-17 at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Ikast Ottosen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Center for Translational Cardiology and Pragmatic Randomized Trials, Herlev and Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Yes